CLINICAL TRIAL: NCT05290194
Title: Multi-target Radiotherapy Combined With PD-1 Monoclonal Antibody and Capecitabine Maintenance Therapy Treating Oligometastatic Nasopharyngeal Carcinoma: a Single-arm, Multicenter, Prospective, Open-label Phase II Clinical Trial
Brief Title: Radiotherapy Combined With PD-1 Monoclonal Antibody and Capecitabine in the Treatment of Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhigang Liu, Chief physicion, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY[2022]LunziNo.(K11-1)
Record Dates: First submitted 2022-03-05; First posted 2022-03-22 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Radiotherapy; PD-1 Inhibitor; Capecitabine; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Immune Checkpoint Inhibitors; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oligometastatic nasopharyngeal carcinoma (Experimental): Patients included are going to receive radiotherapy, chemotherapy and immunotherapy. Radiotherapy includes IMRT and SBRT. IMRT is applied for primary sites and cervical lymph nodes，and SBRT following is applied for oligometastatic sites. PD-1 inhibitors: during the whole trial, intravenous, Q3W; Capecitabine: 650mg, po, bid, following the radiotherapy for a year.
  Interventions: Radiation: SBRT radiotherapy + Conventionally fractionated radiotherapy; Drug: PD-1 inhibitor; Drug: Capecitabine

INTERVENTIONS:
Radiation: SBRT radiotherapy + Conventionally fractionated radiotherapy — Radiotherapy was performed 3-6 weeks after the end of first-line treatment, followed by conventional fractionated radiotherapy of the primary tumor and cervical lymph node metastases, SBRT radiotherapy of distant organ metastases 3-6 weeks later.
Drug: PD-1 inhibitor — Immunotherapy of PD-1 inhibitor is used during the whole time of this trial until subjects were withdrawn from the trial or the trial complete
  Other Names: Immune Checkpoint Inhibitors
Drug: Capecitabine — Capecitabine is treated for patients 3-6 weeks after radiotherapy, which combines with PD-1 inhibitor as the maintenance regimen in the trial.
  Other Names: Xeloda

SUMMARY:
This is a single-arm, multicenter, prospective, open-label phase II clinical trial of multi-target radiotherapy combined with PD-1 monoclonal antibody and capecitabine maintenance therapy treating oligometastatic nasopharyngeal carcinoma, the main purpose of which is to evaluate the efficacy of multi-target radiotherapy combined with PD-1 monoclonal antibody and capecitabine maintenance therapy regimen in treating oligometastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a single-arm, multicenter, prospective, open-label phase II clinical study of multi-target radiotherapy combined with PD-1 monoclonal antibody and capecitabine maintenance therapy for oligometastatic nasopharyngeal carcinoma. Its primary objective is to assess the efficacy, including progression-free survival (PFS), 2-year overall survival (Two-year OS) and progression-free survival (Two-year PFS), overall survival (OS), duration of response (DOR) and safety of multi-target radiotherapy combined with PD-1 monoclonal antibody and capecitabine maintenance therapy in treating oligometastatic nasopharyngeal carcinoma. The secondary objective is to explore the potential genetic biomarkers and clinical therapeutic efficacy evaluation and prediction model of multi-target radiotherapy combined with PD-1 monoclonal antibody and capecitabine maintenance therapy regimen in treating oligometastatic nasopharyngeal carcinoma, providing the evidence of the screening of the potential patients benefiting from the regimen of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was histologically or cytologically diagnosed with nasopharyngeal carcinoma;
2. The patient was newly diagnosed with metastatic nasopharyngeal carcinoma (AJCC eighth edition), and after 4-6 cycles of gemcitabine plus cisplatin combined with PD-1 monoclonal antibody regimen, the efficacy reached more than stable disease;
3. Except for the primary tumor and cervical lymph node metastasis, less than 5 distant organ metastases, and were suitable for SBRT radiotherapy;
4. ECOG PS score 0-2 points;
5. Aged 18-70 years old;
6. Major organ function met the following criteria (14 do not allow the use of any blood components and cell growth factor):

   1. Neutrophil ANC ≥ 2.0 × 10^9/L; platelet count PLT ≥ 100 × 10^9/L; hemoglobin HB ≥ 90 g/L;
   2. Serum albumin ≥ 28 g/L;
   3. Alanine aminotransferase ALT, aspartate aminotransferase AST ≤ 2.5 × ULN; if there is liver metastasis, ALT and AST ≤ 5 × ULN;
   4. Serum creatinine ≤ 1.5 × ULN, Or creatinine clearance ≥ 60 mL/min;
   5. INR ≤ 1.5 × ULN, and APTT ≤ 1.5 × ULN;
7. Life expectancy ≥ 12 weeks;
8. The subject who voluntarily joins the study, sign informed consent, and coordinates with follow-up.

Exclusion Criteria:

1. Recurrent and metastatic nasopharyngeal carcinoma after initial treatment;
2. Patients received previous treatment of primary lesion or metastasis except for the standard first-line regimen (gemcitabine plus cisplatin combined with PD-1 monoclonal antibody regimen), including induction chemotherapy, adjuvant chemotherapy, concurrent chemoradiotherapy, surgery and other treatments;
3. Central nervous system metastastic (confirmed or suspected);
4. Allergy to PD-1 monoclonal antibody or other PD-1 monoantibody; intolerance or allergy to capecitabine; suffering any disease or extrinsic factors affecting oral drugs;
5. Uncontrolled cardiac clinical symptoms or diseases, such as: ① heart failure of NYHA Grade II or higher ; ② unstable angina pectoris; ③ suffering myocardial infarction within 1 year; ④ patients with supraventricular or arrhythmia requiring clinical intervention;
6. Severe infection (CTCAE 5.0 ≥ 2) 4 weeks before the first use of study drugs, such as severe pneumonia, bacteremia, infectious complications requiring hospitalization; baseline chest imaging examination suggests the presence of active pulmonary inflammation; symptoms and signs of infection or the need for oral or intravenous antibiotics (excluding the prophylactic use of antibiotics) 2 weeks before the first use of the study drug;
7. History of other malignancies within 5 years or at the time,but except for cured cutaneous basal cell carcinoma and cervical carcinoma in situ, breast carcinoma in situ, superficial bladder tumors (Ta, Tis and T1) and papillary thyroid cancer as well as other cancers treated more than 3 years before the start of the study;
8. Any of the following conditions is met:

   1. Received any investigational drug before the first use of the study drug;
   2. Participated in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or interventional clinical study at the follow-up time;
   3. Required systemic treatments with corticosteroids (the dose higher than the equivalent dose of 10 mg prednisone per day) or other immunosuppressive agents 2 weeks before the first use of the study drug, except for local inflammation and prevention of allergy and nausea and vomiting. In the absence of active autoimmune disease, inhaled or topical steroids and adrenocorticotropic hormone replacement at doses greater than 10 mg daily in prednisone efficacy dose are allowed;
   4. Received anti-tumor vaccines or vaccinated live vaccines 4 weeks before the first dose of study drug;
   5. Underwent excessive surgery or severe trauma 4 weeks before the first use of study drug;
9. Patients had active autoimmune diseases and a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes) in the past 2 years; patients who did not require any intervention after adulthood are allowed;
10. History of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation and bone marrow transplantation;
11. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection 1 year ago but without regular treatment;
12. Patients with active hepatitis (HBV ≥ 2000 IU/ml or HBV DNA ≥ 10000/ml), or hepatitis C (hepatitis C antibody positive, and HCV-RNA ≥ 1000/ml);
13. Patients with coagulation abnormalities (PT > 16s, APTT > 43s, TT > 21s, Fbg < 2 g/L), bleeding tendency or receiving thrombolytic or anticoagulant therapy; or patients with previous severe bleeding (bleeding > 30ml within 3 months), hemoptysis (bleeding > 5ml within 4 weeks) within 12 months due to thromboembolic events (including stroke events and/or transient ischemic attack);
14. Uncontrolled hypertension (systolic blood pressure > 140 mmHg, or diastolic blood pressure > 90 mmHg); coronary heart disease, arrhythmia ≥ grade II (including QTc prolongation, male > 450 ms, female > 470 ms) and heart failure;
15. Urine protein ≥ + +, or 24 hour urine protein ≥ 1.0 g;
16. Current diarrhea-related diseases (e.g., ulcerative colitis, Crohn's disease, chronic diarrhea, etc.);
17. Known history of psychotropic drug abuse, alcoholism and drug abuse; or current history of antiepileptic drug use;
18. Pregnant or lactating;
19. Patients considered unsuitable for inclusion by the investigator as assessed by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 2 years
  The time between enrollment and progression(in any way) or death (for any reason)

SECONDARY OUTCOMES:
Overall survival | 2years
  Time from randomization to death (for any reason)
Duration of response | 2 yaers
  Time from the first evaluation of the tumor as CR or PR to the first evaluation as PD or death from any cause

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 years
  The incidence of adverse events (≥Grade 2，CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang MD Liu, PhD, Principal Investigator — Fifth Affilliated Hospital of Sun Yat-sen University
Locations (1):
- Fifth Affilliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided